CLINICAL TRIAL: NCT04298801
Title: Does the Implementation of Nurse-driven HIV Screening for Key Populations in the Emergency Departments Limit Undiagnosed Infections in the Paris Metropolitan Area?
Brief Title: Does the Implementation of Nurse-driven HIV Screening for Key Populations in the Emergency Departments Limit Undiagnosed Infections in the Paris Metropolitan Area? DEPIST Trial (ANRS 14055)
Acronym: DEPIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: APHP190502; 2019-A02364-53 (Other: ANSM); ANRS 14055 (Other: ANRS)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Hiv; Nurse's Role
Keywords: Emergency service, Hospital; HIV; Mass screening; Nurses; Prevention and control; Key populations; Targeted screening
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-driven HIV screening for key populations+UD (Experimental): Nurse-driven HIV screening for key populations combined with usual physician-directed diagnostic testing (UD)
  Interventions: Procedure: Nurse-driven HIV screening for key populations combined with usual physician-directed diagnostic testing; Other: Physician-directed diagnostic testing
- Physician-directed diagnostic testing alone (Active Comparator)
  Interventions: Other: Physician-directed diagnostic testing

INTERVENTIONS:
Procedure: Nurse-driven HIV screening for key populations combined with usual physician-directed diagnostic testing — A self-administered questionnaire on HIV exposure factors will be offered to all patients of ages 18-64 able to complete it. This questionnaire will be available in a paper-based format, electronic format on the patient phone or can be conducted verbally by the nurse. According to the answers, the nurses will suggest performing a rapid test to patients belonging to key populations. A finger-stick rapid HIV test will be performed and results will be disclosed by the nurse assisted by a physician if necessary.
  If needed, a follow-up visit with an infectious disease specialist will be scheduled within 72 hours.
  Arms: Nurse-driven HIV screening for key populations+UD
Other: Physician-directed diagnostic testing — Throughout the intervention, physicians will prescribe HIV tests to patients with HIV-related symptoms, following usual practice.

SUMMARY:
In France, 40% of newly diagnosed HIV infections are concentrated in the Paris metropolitan area.

Two key populations are mainly concerned: persons born in a foreign country and men who have sex with men. The randomized trial ANRS DICI-VIH (2014-2015) showed that nurse-driven HIV screening for key populations, supported by research staff, in 8 emergency departments (EDs) of the region, was effective in addition to diagnostic testing. The strategy advocated by the WHO and the recent French recommendations support the proposal of screening for key populations in the EDs. Thus, it is important to evaluate the impact and the feasibility of the implementation of this strategy on a large scale.

The aim is to evaluate the impact of a wide implementation of nurse-driven HIV screening by rapid test in key populations combined with usual physician-directed diagnostic testing (intervention strategy) compared to diagnostic testing alone (control strategy) in the usual practice of the EDs.

The strategies will be compared during two periods in 18 EDs of Paris metropolitan area following a stepped-wedge cluster randomized trial.

During intervention period, nurses will suggest performing an HIV rapid test to patients belonging to key populations according to the answers to a self-administered questionnaire.

DETAILED DESCRIPTION:
Background:

In France, 40% of newly diagnosed HIV infections are concentrated in the Paris metropolitan area.

Two key populations are mainly concerned: persons born in a foreign country and men who have sex with men. The randomized trial ANRS DICI-VIH (2014-2015) showed that nurse-driven HIV screening for key populations, supported by research staff, in 8 emergency departments (EDs) of the region, was effective in addition to diagnostic testing. The strategy advocated by the WHO and the recent French recommendations of the National Health Authority (HAS) and expert group support the proposal of screening for key populations in the EDs. Thus, it is important to evaluate the impact and the feasibility of the implementation of this strategy on a large scale in a context where local institutions are taking initiatives to curb the epidemic ("Pour une Ile-de-France sans sida", "Vers Paris sans sida").

Our hypothesis is that nurse-driven HIV screening for key populations can be integrated to the consultants' care pathway as usual practice of the ED and assured over the long term in the Paris metropolitan area; this strategy combined with physician-directed diagnostic testing could reduce undiagnosed infections and help control the epidemic.

Primary objective:

The primary objective is to evaluate the impact of a wide implementation of nurse-driven HIV screening by rapid test in key populations combined with usual physician-directed diagnostic testing (intervention strategy) compared to diagnostic testing alone (control strategy) in the usual practice of the EDs.

Patients aged 18 to 64 years and visiting a participating ED for reasons other than a potential exposure to HIV within less than 48 hours will be included.

The primary outcome is the proportion of new HIV diagnoses among included patients.

Secondary objectives are to :

* evaluate the feasibility of nurse-driven screening and its long-term implementation,
* evaluate the effectiveness of the screening process used by the caregivers, particularly the use of an electronic questionnaire, and by the patients as well as the acceptability,
* compare newly diagnosed HIV+ patients in the two groups in terms of :

  1. linkage to follow up care,
  2. proportions of patients who had a CD4 cell count greater or equal to 500 or 350 cells/µL and no HIV-related symptoms and proportions of patients with acute HIV infection.
* estimate through modelling the number of new HIV diagnoses for different levels of coverage of the screening strategy in the Paris metropolitan area.

Methods The strategies will be compared in 18 EDs of Paris metropolitan area during two periods. The start of the intervention strategy will be randomly allocated for each ED following a stepped-wedge cluster randomized trial.

EDs are selected according to the proportion of patients belonging to key populations in the patients they receive (data from two previous studies).

During intervention period, nurses will suggest performing an HIV rapid test to patients belonging to key populations according to the answers to a self-administered questionnaire.

The intervention period will last 3 to 11 months and the control period 0 to 8 months. Patients will participate up to 1 month if a follow-up is needed.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18 to 64 years and visiting a participating ED for reasons other than a potential exposure to HIV within less than 48 hours

Exclusion Criteria:

- Not applicable

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 487000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of new HIV diagnoses among included patients. | At the end of the expected total duration of the inclusion period: 11 months in each ED

SECONDARY OUTCOMES:
Feasibility of the screening strategy and its implementation | At the end of the expected total duration of the inclusion period: 11 months in each ED
  Feasibility of the screening strategy and its implementation based on:
  * proportion of distributed and completed self-administered questionnaires among the patients included and among the patients able to participate who were not known to be HIV positive,
  * the proportion of rapid tests offered by nurses among patients belonging to key populations,
  * the proportion of patients screened by nurses among patients who were offered a rapid test and among patients belonging to high-risk groups .
Effectiveness of the screening processes used by the caregivers, particularly the integration of the electronic questionnaire, and used by the patients as well as acceptability | At the end of the expected total duration of the inclusion period: 11 months in each ED
Proportions of patients with a new diagnosis | At the end of the expected total duration of the inclusion period: 11 months in each ED
  Proportions of patients with a new diagnosis who had:
  * a follow up visit with an infectious disease specialist within 1 month,
  * a CD4 cell count greater or equal to 500 or 350/µL and no HIV-related symptoms,
  * an acute HIV infection.
Estimation through modelling of the number of new HIV diagnoses for different levels of coverage of the screening strategy in the Paris metropolitan area. | At the end of the expected total duration of the inclusion period: 11 months in each ED

CONTACTS AND LOCATIONS:
Overall Officials: judith LEBLANC, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided